CLINICAL TRIAL: NCT04576845
Title: The Effect of Early Childhood Cow's Milk Allergy Elimination Diet on Eating Behaviors, Nutrition, and Growth Status at Age 2-6
Brief Title: The Effect of Early Childhood Cow's Milk Allergy Elimination Diet on Eating Behaviors, Nutrition, and Growth Status
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nazlı ERCAN, Pediatric Allergy and Immunology specialist, MD, Saglik Bilimleri Universitesi
Other Study IDs: NazliKubra2020
Record Dates: First submitted 2020-09-17; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Nutrient Deficiency; Eating Behavior; Cow Milk Allergy; Growth Disorders
Keywords: Cow's Milk Protein Allergy (CMA); Children's Eating Behavior Questionnaire (CEBQ); Elimination diet; Eating behavior; Food fussiness
MeSH Terms: conditions — Feeding Behavior; Milk Hypersensitivity; Growth Disorders; Food Fussiness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: The study will be performed on Caucasian origin children who are among 2 to 6 years of age. The study group will be composed of children (n=31) who had CMA (Ig E-mediated and/or non-Ig E-mediated and/or mixed type) proved with oral food challenge tests in their early childhood (in ages of 0-2). The inclusion criteria to the study group will be to undergo a Cow's milk elimination (CME) diet or took a hypoallergenic formula in 0-2 years of age for at least 3 months or longer due to CMA allergy and improved afterward, and/or to eliminate other nutrients (e.g., eggs, potatoes, wheat flour, soybean, etc.) other than cow's milk between the ages of 0-2 for at least 3 months or longer, and/or to add these nutrients back to their diet in the last 3 months, and/or not receiving hypoallergenic formula for the last 3 months, not to be on the CME diet at present. Thus, no children in the study and control groups will be on a dietary restriction during the study.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The children's eating behavior will be evaluated with Turkish validated Children's Eating Behavior Questionnaire - (CEBQ) by interviewing mothers face to face. The CEBQ is a Likert type, parent-report rating scale measuring the variation in eating behavior in children. The CEBQ consists of 35 items comprising eight subscales, each containing 3 to 6 items. Parents will be asked to rate their child's eating behavior on a five-point scale (never, rarely, sometimes, often, always; 1-5, respectively).
  Other Names: The children's eating behavior will be evaluated with Turkish validated Children's Eating Behavior Questionnaire - (CEBQ)

SUMMARY:
Cow's milk allergy (CMA) is the most common Food Allergy (FA) in children, and the essential strategy in prevention is avoiding the allergens that may cause potentially life-threatening reactions.

The primary developmental task of early childhood is the creation of healthy eating habits. The diagnosis of FA in this period can lead to permanent changes in the life of the child and her family. In early childhood, parents are often responsible for all aspects of FA management because children are too young to understand the complexity of avoiding allergens. Children often do not have the skills to implement FA management. Parents are advised to follow a special weaning diet, avoiding any type of cow's milk, usually at least 1 year old. However, depending on the clinical improvement, it can be recommended to continue this exclusion diet for much longer. Thus, many children have to exclude a large group of food from their diets, which is critical for their growth, development, and eating habits. This may raise mealtime behavioral anxiety in a child with a FA.

Eating behavioral anxieties are also very common in healthy, typically developing children. Even 25% to 45% of normally developing children's parents report concerns about their child's nutritional and mealtime behaviors, including the destructive child behaviors (eg., refusal of foods, food selectivity, and getting off the table).

In children with food allergies, monitoring long-term growth after the diet is another important issue. Growth problems were reported in 21% of children with FA diagnosed with malnutrition. Most studies focused on the effect of changes in eating behavior on growth during an elimination diet or in short term intervals. Its long-term effects have only been analyzed in a few studies. We aimed to investigate the eating behaviors, nutritional status, and growth of young children (ages of 2 to 6) who had a strict diet due to CMA in early childhood (ages of 0-2).

DETAILED DESCRIPTION:
Study Design The study is planned to be a cross-sectional, case-control study and it will be carried out between October 2020 and November 2020 in our tertiary care center (university hospital located in Ankara, Turkey). The study will be conducted with the collaboration of the departments of Pediatric Immunology and Allergy and Nutrition and Dietetics. The study was approved by our University ethics committee (2011- KAEK-19) with the decision number of 108/2019. The children eligible for the study group will be enrolled from the pediatric allergy and immunology outpatient unit. The control group children will be selected from the health visitor clinics of Pediatrics. The patient informed consent form will be obtained from all children's parents at the beginning of the study.The study will be performed on Caucasian origin children who are among 2 to 6 years of age. The study group will be composed of children (n=31) who had CMA (Ig E-mediated and/or non-Ig E-mediated and/or mixed type) proved with oral food challenge tests in their early childhood (in ages of 0-2). The control group (n=31) will include healthy children who had never been on a diet throughout their lives. No children in the study and control groups will be on a dietary restriction during the study. The inclusion and the exclusion criteria are given in detail at the space for eligibility.

Data collection The children's eating behavior will be evaluated with Turkish validated Children's Eating Behavior Questionnaire - (CEBQ) by interviewing mothers face to face. The CEBQ is a Likert type, parent-report rating scale measuring the variation in eating behavior in children. The CEBQ consists of 35 items comprising eight subscales, each containing 3 to 6 items. Parents were asked to rate their child's eating behavior on a five-point scale (never, rarely, sometimes, often, always; 1-5, respectively).

The 8 subscales of CEBQ and their interpretation are: The sub-scales Satiety Responsiveness (SR) (i.e., "My child has a big appetite", 7 items), Slowness in Eating (SE) (i.e., "My child eats slowly", 4 items), Emotional Undereating (EUE) (i.e., "My child eats less when she/he is tired", 4 items), and Food Fussiness (FF) (i.e., "My child refuses new foods at first", 3 items) assess "food avoidance" (i.e., increased internal satiety and avoidance of eating), while the sub-scales Food Responsiveness (FR) (i.e., "My child is always asking for food", 5 items), Enjoyment of Food (EF) (i.e., "My child loves food", 5 items), Desire to Drink (DD) (i.e., "My child is always asking for a drink", 3 items), and Emotional Overeating (EOE) (i.e., "My child eats more when worried", 4 items) assess "food approach" (i.e., high responsiveness to food). Higher scores indicate a stronger display of food approach or food avoidance (except FF) behavior. In the Turkish version of the CEBQ, a lower score for FF means a stronger display for fussy eating. Therefore, while calculating the food avoidance total score, reversed items of FF were summed with SR, SE, and EUE. The food approach total score will be calculated by the summation of FR, EF, DD, and EOE.

Another questionnaire that will be conducted with the mothers will be to discuss their socio-demographic characteristics. Three days' food record will be obtained from each mother (2 weekdays and 1 weekend day). On the same days, the food consumed by children at school will be recorded by the teachers, and consumption registration forms will be combined at the end of three days. Portion sizes and volumes will be estimated with a portion size picture book, including 120 photographs of foods, each with 3-5 different portion sizes. In addition, each serves of participants will be confirmed with the pictures taken by the parents that will show the plates of their children before and after each meal. Only the forms accurately registered will be evaluated. BeBiS software version 7.2 will be used to calculate the daily intake of energy, macronutrients, micronutrients, and dairy products. The Nutrition Guide will be assessed the adequacy of children's nutrient intake for Turkey according to age and gender. The same researcher will take the body weights (kg) and height (cm) of the children with the same method, previously described by the World Health Organization (WHO) using the same measuring instruments. Measurements will be performed using the standardized Conformité Européene marked scales and stadiometers [A baby scale (Testut, Paris) will be used for infants weighing <15 kg and an electronic scale (Seca, Hamburg, Germany) will be used for children weighing >15 kg. Seca 213 and infantometer will be used for measuring participants' height]. Scale and stadiometer are routinely calibrated in our hospital according to rules of quality. Body Mass Index (BMI) will be calculated with the formula kg/m2. The anthropometric (height-for-age [HFA], weight-for-age [WFA], and body mass index-for-age [BMI]) measurements will be evaluated according to the Z-score using the WHO ANTHRO program (Version 3.2.2, January 2011) and WHO ANTHRO Plus Software (WHO, 2009b) [Z-score = Patient's value - Average value / Standard Deviation (SD)]. The Z-score (SDS) in the average child by age will be "0". Values between +2 SD and - 2 SD will be considered normal upper and lower limits.

Primarily, we will compare the eating behavior of children who had a strict CME diet due to CMA in early childhood with healthy children. Secondarily, we will evaluate the effects of children's eating behavior on participants' nutritional status and anthropometric measurements.

ELIGIBILITY:
The inclusion criteria to the study group will be as follows;

1. to undergo a Cow's milk elimination (CME) diet or took a hypoallergenic formula in 0-2 years of age for at least 3 months or longer due to CMA allergy
2. improvement of CMA after receiving CME diet,
3. to eliminate other nutrients (e.g., eggs, potatoes, wheat flour, soybean, etc.) other than cow's milk between the ages of 0-2 for at least 3 months or longer,
4. to add other nutrients (as mentioned in criterion 3) back to their diet in the last 3 months,
5. not receiving hypoallergenic formula for the last 3 months,
6. not to be on the CME diet at present.

The exclusion criteria from enrollment to the study will be as follows;

1. Children with any disease that may affect eating behavior, nutritional status, and growth.
2. The children with a diagnosis of a disease mentioned below will be excluded from the study.

   1. Children with a diagnosis of chronic infection / inflammatory diseases,
   2. cystic fibrosis,
   3. congenital heart disease,
   4. chronic kidney failure,
   5. diabetes,
   6. gastroesophageal reflux,
   7. dysfunction of swallowing,
   8. anatomical, cognitive and/or impairment of speech,
   9. autoimmune diseases (SLE, RA, thyroid, etc.),
   10. congenital genetic diseases,
   11. immune deficiency,
   12. autism,
   13. attention deficit hyperactivity,
   14. manic-depressive disorders.

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: The children eligible for the study group will be enrolled from the pediatric allergy and immunology outpatient unit. The control group children will be selected from the health visitor clinics of Pediatrics. All children will be enrolled in the study will be Caucasian origin between 2 to 6 years of age. The study group will be composed of children (n=31) who had CMA (Ig E-mediated and/or non-Ig E-mediated and/or mixed type) proved by oral food challenge test in their early childhood (in ages of 0-2). The control group (n=31) will include healthy children who had never been on a diet throughout their lives.
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2020-10-12 (Estimated); Primary Completion 2020-11-13 (Estimated); Study Completion 2020-11-13 (Estimated)

PRIMARY OUTCOMES:
Eating behavior will be evaluated by CEBQ scoring system. | One day
  The 8 subscales of CEBQ and their interpretation are: The sub-scales Satiety Responsiveness (SR) (7 items), Slowness in Eating (SE) (4 items), Emotional Under Eating (EUE) (4 items), and Food Fussiness (FF) (3 items) assess "food avoidance", while the sub-scales Food Responsiveness (FR) (5 items), Enjoyment of Food (EF) (5 items), Desire to Drink (DD) (3 items), and Emotional Overeating (EOE) (4 items) assess "food approach". Higher scores indicate a stronger display of food approach or food avoidance (except FF) behavior. In the Turkish version of the CEBQ, a lower score for FF means a stronger display for fussy eating. Therefore, while calculating the food avoidance total score, reversed items of FF were summed with SR, SE, and EUE. The food approach total score will be calculated by the summation of FR, EF, DD, and EOE.

SECONDARY OUTCOMES:
BeBiS software version 7.2 will be used to calculate the daily intake of energy, macronutrients, micronutrients, and dairy products. | (2 weekdays and 1 weekend day).
  Three days' food record will be obtained from each mother (2 weekdays and 1 weekend day). On the same days, the food consumed by children at school will be recorded by the teachers, and consumption registration forms will be combined at the end of three days. Portion sizes and volumes will be estimated with a portion size picture book, including 120 photographs of foods, each with 3-5 different portion sizes. Each serves of participants will be confirmed with the pictures taken by the parents showing children's plates before and after each meal. Only the forms accurately registered are planned to be evaluated. The adequacy of children's nutrient intake will be assessed with the Nutrition Guide for Turkey according to age and gender.
The anthropometric evaluation of children respecting body weight. | One day
  The same researcher will take the body weights (in kilograms = kg) of the children with the method described by the World Health Organization (WHO) using the same measuring instruments. Measurements will be performed using the standardized Conformité Européene marked scales and stadiometers. A baby scale (Testut, Paris) will be used for infants weighing <15 kg, and an electronic scale (Seca, Hamburg, Germany) will be used for children weighing >15 kg.
The anthropometric evaluation of children respecting height. | One day
  The same researcher will take the height (in centimeters = cm) of the children with the method described by the World Health Organization (WHO) using the same measuring instruments. Measurements will be performed using the standardized Conformité Européene marked scales and stadiometers. Seca 213 and infantometer will be used for measuring participants' height.
The anthropometric evaluation of children with calculation of BMI. | One day
  The measured weight (in kilograms) and height (in centimeters; The unit conversion to meters will be performed by dividing cm to 100). BMI of children will be calculated with the formula kg/m2.
Z-score calculations of all participants using WHO ANTHRO program. | One day
  The anthropometric (height-for-age [HFA], weight-for-age [WFA], and body mass index-for-age [BMI]) measurements will be evaluated according to the Z-score using the WHO ANTHRO program and WHO ANTHRO Plus Software.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maslin K, Grundy J, Glasbey G, Dean T, Arshad SH, Grimshaw K, Oliver E, Roberts G, Venter C. Cows' milk exclusion diet during infancy: Is there a long-term effect on children's eating behaviour and food preferences? Pediatr Allergy Immunol. 2016 Mar;27(2):141-6. doi: 10.1111/pai.12513. Epub 2016 Jan 21. PMID 26592369
- [Result] Meyer R, Rommel N, Van Oudenhove L, Fleming C, Dziubak R, Shah N. Feeding difficulties in children with food protein-induced gastrointestinal allergies. J Gastroenterol Hepatol. 2014 Oct;29(10):1764-9. doi: 10.1111/jgh.12593. PMID 24720353
- [Result] Mukkada VA, Haas A, Maune NC, Capocelli KE, Henry M, Gilman N, Petersburg S, Moore W, Lovell MA, Fleischer DM, Furuta GT, Atkins D. Feeding dysfunction in children with eosinophilic gastrointestinal diseases. Pediatrics. 2010 Sep;126(3):e672-7. doi: 10.1542/peds.2009-2227. Epub 2010 Aug 9. PMID 20696733
- [Derived] Ercan N, Tel Adiguzel K. Effect of early childhood cow's milk elimination diet on eating behaviours, nutrition and growth status at age 2-6 years. J Hum Nutr Diet. 2022 Apr;35(2):300-309. doi: 10.1111/jhn.12914. Epub 2021 Jun 16. PMID 33974304